CLINICAL TRIAL: NCT00237822
Title: Increasing Treatment Adherence in Co-Occurring Disorders
Brief Title: Increasing Treatment Adherence in Co-Occurring Psychiatric and Drug Use Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: K23DA015144 (NIH); K23DA015144 (NIH)
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2005-10

CONDITIONS: Diagnosis, Dual (Psychiatry); Psychiatric Diagnosis; Drug Use Disorders
Keywords: Treatment Adherence; Co-Occurring Disorders; Motivational Enhancement Therapy; Contingency Management; MEMS Caps
MeSH Terms: conditions — Disease; Mental Disorders; Substance-Related Disorders; Treatment Adherence and Compliance | interventions — Motivational Interviewing

INTERVENTIONS:
Behavioral: Adherence Feedback (AF)
Behavioral: AF + Contingency Management (AF + CM)
Behavioral: AF + Motivational Enhancement Therapy (AF + MET)

SUMMARY:
The investigators are proposing a study of treatment adherence in co-occurring psychiatric and drug use disorders (COD). The proposed study uses a 3-cell/condition design, within which 75 adult outpatients with co-occurring psychiatric disorders and drug abuse/dependence (CODDA) will be randomly assigned to one of the following brief, 8-week, manual-guided interventions following a 2-week "Assessment Only" baseline period:

1. Adherence Feedback (AF); this condition will entail weekly, 20-25 minute sessions of AF, which is a procedure that represents a technological advancement developed by Cramer et al. (1989, 1995, and 1999) and is based on the use of adherence data from the microelectronic monitor in Medication Event Monitoring System (MEMS) caps,
2. AF + Contingency Management (AF + CM); in this condition, participants will receive AF, as described above, PLUS contingency management. CM is based on the behavioral learning theory, which suggests that the occurrence of a behavior is increased as a function of the rate at which it is positively reinforced or rewarded, or
3. AF + Motivational Enhancement Therapy (AF + MET); in this condition, patients will receive AF, as described above, PLUS motivational enhancement therapy. MET is based on the idea that an effective way to motivate behavior change is to assist patients in clarifying their ambivalence (i.e., reasons for and against changing/adhering), utilizing a series of strategies based on client-centered psychotherapy, self-efficacy theory, and social psychology.

The study will allow the evaluation of three hypotheses:

1. AF + MET is superior to AF + CM,
2. AF + MET is superior to AF alone, and
3. AF + CM is superior to AF alone.

Primary outcome measures are:

1. rates of adherence to medication (i.e., selective serotonin reuptake inhibitors or SSRIs), as measured by MEMS caps and self-report,
2. rates of counseling attendance, and
3. reductions in illicit drug use, including achievement of abstinence, as assessed by twice-weekly urine toxicology tests and self-report.

Secondary outcomes include reductions in psychiatric symptomatology and rates of re-hospitalization. The investigators will also evaluate the relationship between adherence and primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Currently being treated with any class of psychotropic medication
* Have used illicit drugs or abused prescription drugs within the past year
* Are not adhering completely to their medication

Exclusion Criteria:

* Current major depressive episode
* Active suicidal/homicidal ideation/intent
* Current manic episode
* Visiting nurse or living in a facility that distributed medications

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2003-09; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Treatment adherence

SECONDARY OUTCOMES:
Drug use
Depression

CONTACTS AND LOCATIONS:
Overall Officials: Michael V. Pantalon, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University Substance Abuse Center, New Haven, Connecticut, United States